CLINICAL TRIAL: NCT01100476
Title: Single-center, Post Market, Prospective, Consecutive, Single-arm Study Compared to Historical Control (Diagnostic Arm of the Mynx 6/7F Study)
Brief Title: Mynx M5 One Hour Ambulation Study
Acronym: Mynx
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cardiovascular Associates of the Delaware Valley (Other)
Collaborators: AccessClosure, Inc. (Industry)
Responsible Party: Principal Investigator, Vijayendra K. Verma, MD, Principal Investigator, Cardiovascular Associates of the Delaware Valley
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010 - M5
Record Dates: First submitted 2010-04-05; First posted 2010-04-09 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Angiography
Keywords: Closure Device; endovascular procedures; sealing femoral arterial access; Mynx M5
MeSH Terms: interventions — Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Endovascular Diagnostic Procedures — Patients underwent a percutaneous diagnostic procedure utilizing a 5F procedural sheath in the common femoral artery
  Other Names: Angiography

SUMMARY:
The Mynx Vascular Closure Device (Mynx M5) is a sponge-like material used to close the hole in the artery after patients undergo a diagnostic endovascular procedures

DETAILED DESCRIPTION:
Key Inclusion:

1. Patients >18 yrs of age
2. Patient underwent a percutaneous diagnostic procedure utilizing a 5F procedural sheath via the common femoral artery.
3. Patient is able to ambulate (routinely walk 6 meters or 20 feet without assistance for any reason) as assessed by investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years of age
* Patient underwent a percutaneous diagnostic procedure utilizing a 5F procedural sheath in the common femoral artery
* Patient has been informed and understands the nature of the study and provides written INformed COnsent approved by the appropriate Institutional Review Board (IRB) prior to enrollment
* Patient is able to ambulate (routinely walk 6 meters or 20 feet without assistance for any reason) as assessed by the investigator

Exclusion Criteria:

Pre-Procedure Exclusion Criteria

* Patient had a prior surgical procedure, PTA, stent placement, or vascular graft in the common femoral artery
* Patient has a bleeding disorder such as thrombocytopenia
* Patient has uncontrolled hypertension
* Patient is morbidly obese (BMI >40 kg/m2
* Patient is pregnant or lactating
* Patient has a documented INR >1.5 or patients currently receiving glycoprotein IIb/IIIa platelet inhibitor
* Patient has a known severe allergy to contrast medium
* Patient has a known allergy to PEG
* Patient is unable to ambulate at one hour secondary to a co-morbid condition
* Patient is know to require an extended hospitalization or re-hospitalization (e.g.patient is undergoing coronary artery bypass graft (CABG) surgery) or patient is scheduled to have a CABG surgery <30 days following the procedure

Intra-Procedure Exclusion Criteria

* Common femoral artery is <5mm in diameter
* Patient with clinically significant peripheral vascular disease in the vicinity of the puncture
* Puncture site is located above the most inferior border of the inferior epigastric artery (IEA) and/or above the inguinal ligament based upon bony landmarks
* Patient has a posterior puncture or multiple punctures in an attempt to gain access
* Patient has an ipsilateral venous sheath
* Patient has a pre-existing arterial bleed/extravasation identified on pre-procedure femoral arteriogram, hematoma, pseudoaneurysm or arteriovenous fistula present prior to sheath removal
* Patient has intra-procedural bleeding around the access site prior to sheath removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety & Tolerability | Enrollment approx for 4 months
  To assess safety and tolerability of participants ambulating within one hour of placement of the Mynx M5 Closure Device. Participants will be assessed for adverse event occurrence for 30 +/-7 days.

SECONDARY OUTCOMES:
Device success | 30 +/- 7days
  Assess device success, time to dischargeability, major and minor complications in all patients enrolled in the study

CONTACTS AND LOCATIONS:
Overall Officials: Vijay K Verma, MD, Principal Investigator — Cardiovascular Associates of the Delaware Valley; Mary F Kinder, RN, BSN, Study Director — Cardiovascular Associates of the Delaware Valley
Locations (1):
- Our Lady of Lourdes Medical Center, Camden, New Jersey, United States